CLINICAL TRIAL: NCT00157885
Title: A Randomized Trial to Compare the Efficacy of Artekin and Amodiaquine Plus Artesunate for the Treatment of Acute Falciparum and Vivax Malaria in Timika, Papua
Brief Title: A Randomised Trial of Artekin and Artesunate & Amodiaquine for Uncomplicated Malaria in Timika, Papua, Indonesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other); Wellcome Trust (Other); National Health and Medical Research Council, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Timika_AMT; Welcome Trust ME028458MES
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-06-26 (Estimated); Status verified 2006-06

CONDITIONS: Malaria, Falciparum; Malaria, Vivax
Keywords: Falciparum; Vivax; Papua; Amodiaquine; Artekin; Artemisinin Combination Therapy; Dihydroartemisinin; Piperaquine; Lumefantrine; Artemether
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax | interventions — Amodiaquine; Artesunate

INTERVENTIONS:
Drug: Amodiaquine plus artesunate; Artekin

SUMMARY:
The primary aim of the comparative trial is to assess the relative safety and efficacy of two artemisinin containing regimens: amodiaquine plus artesunate (AAQ) and artekin both administered once daily for 3 days.

DETAILED DESCRIPTION:
With the emergence of species of multi drug resistant P.falciparum across the archipelago the Indonesian Centre for Disease Control (CDC) now recommends amodiaquine plus artesunate in areas of high chloroquine and sulfadoxine-pyrimethamine resistant strains of P. falciparum. High levels of chloroquine resistance to P.vivax has also emerged in the eastern provinces.

This trial sets out to assess the efficacy of artekin and amodiaquine plus artesunate and artekin against both P.falciparum and P. vivax.

and their safety profiles.

Patients who present to an established rural outpatient clinic in Timika, Papua with symptoms of acute, uncomplicated infection with P. falciparum, P.vivax or both species, will after laboratory confirmation of the diagnosis and having given informed consent to participate in the trial, be enrolled in the study. Patients will be treated as out-patients and then seen daily for the first week until aparasitaemic and thereafter at weekly visits to the clinic.

The data used from this trial will be used to make a public health decision to determine a suitable alternative first line antimalarial in the Timika region. In order to ensure that the data gathered will be relevant to the clinical setting in which the drugs will be used, drug administration of medication will be deliberately designed to mimic conditions that will be experienced with widespread deployment (eg once daily supervision).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least one 1year of age and weighing more than 5kg.
* Microscopic confirmation of P. falciparum and /or P.vivax infection (any parasitaemia).
* Fever (axillary temperature >37.5oC) or history of fever in the last 48 hours.
* Able to participate in the trial and comply with the clinical trial protocol
* Written informed consent to participate in trial; verbal consent in presence of literate witness is required for illiterate patients, and written consent from parents/guardian for children below age of consent

Exclusion Criteria:

* Pregnancy or lactation
* Inability to tolerate oral treatment
* Signs/symptoms indicative of severe/complicated malaria or warning signs requiring parenteral treatment
* Known hypersensitivity or allergy to artemisinin derivatives
* Serious underlying disease (cardiac, renal or hepatic)
* Parasitaemia >4%

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2005-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Overall day 42 cure rate (incorporating early and late treatment failures)

SECONDARY OUTCOMES:
Day 42 P.falciparum cure rate corrected for reinfection by PCR genotyping
Day 42 P.vivax cure rate
Overall day 28 cure rate for P.falciparum
Proportion of patients aparasitaemic on Days 1 and 2
Haematological recovery
Gametocyte Carriage during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ric N Price, MD, Principal Investigator — Menzies School of Health Research; Emiliana Tjitra, Principal Investigator — National Institute of Health Research and Development, Jakarta, Indonesia
Locations (1):
- SP9 & SP12 Public Health & Malaria Control Clinics, Timika, Special Region of Papua, Indonesia